CLINICAL TRIAL: NCT02372851
Title: Assessing the Effectiveness of a Point-of-use Water Filter Technology as an Arsenic Mitigation Strategy in West Bengal
Brief Title: Assessing the Effectiveness of a Water Filter Technology as an Arsenic Mitigation Strategy in West Bengal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Kalyani (Unknown); KIIT University (Unknown); Hindustan Unilever Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LondonSHTM
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2015-09

CONDITIONS: Total Urinary Arsenic; Total Arsenic in Water; Diarrhoeal Disease
Keywords: Arsenic; Household water treatment; Point of use water treatment; Water Quality; Total Urinary Arsenic; West Bengal; Thermotolerant coliforms; Compliance; Diarrhoea
MeSH Terms: conditions — Patient Compliance; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pureit As+ Filter (Active Comparator): Each household will receive one water filter and a replacement battery for free during distribution. The intervention will be distributed door-to-door by the implementation team. Households will be trained on use and maintenance of the device according to the manufacturer's instructions. Households will be advised to drink exclusively from the water filter and to carry water with them if attending school or work. Households will also be advised to clean and cook their rice with filtered water only.
  Interventions: Device: Pureit As+ Filter
- Control arm (No Intervention): The control arm will be advised to continue with their traditional drinking water and cooking practices. The control arm will receive the intervention at the end of the study period.

INTERVENTIONS:
Device: Pureit As+ Filter — The Pureit As+ water filter has been developed to effectively remove arsenic (both arsenite and arsenate) from over 300 µg/L to less than 10 µg/L in addition to removing microbial contamination (Institution of Public Health Engineers, 2011). It has an end-of-life indicator and consumables that do not re-contaminate the environment when disposed (Institution of Public Health Engineers, 2011). The technology requires no electricity, but only the replacement of the battery after 1000 L of water filtered (approximately 100 days based on a family of five drinking 2 L/day).
  Arms: Pureit As+ Filter

SUMMARY:
The purpose of this study is to determine whether the use of a point-of-use water filtration technology can reduce the Arsenic content in drinking water and reduce the Arsenic body burden.

DETAILED DESCRIPTION:
The Unilever Pureit As+ filter will be assessed for chemical and microbiological performance and health impact using a parallel, household-randomised controlled trial (RCT) design over a four-month follow-up period.

This study will follow an open (non-blinded) design because filtration technologies are particularly challenging to blinding (Boisson et al., 2010). Equal randomisation will be applied (i.e. 1:1). Randomisation will be undertaken through a lottery organised in each participating village.

The study will be undertaken in two phases; an initial phase will involve a baseline survey in the identified affected communities. Those households identified as eligible during the baseline survey will then be randomised into the intervention or control group and the intervention will then be distributed. After a 2-4 week adaptation period, control and intervention arms will be followed at monthly visits for a period of four months.

The baseline study will collect information on demographics, sanitation facilities, hygiene practices, drinking water sources and treatment practices, diet of household members, knowledge of arsenic contamination and arsenicosis, and other factors that could potentially impact the outcomes of interest. Additionally, data on behavioural factors that have been observed to be associated with Household Water Treatment (HWT) use will be collected to predict intervention use in the intervention arm. During the baseline survey, water samples of source water and stored drinking water will be collected and tested for total thermotolerant coliforms (TTC) and total arsenic concentration. The female head of the household will be invited to provide a sample of urine for total urinary arsenic testing. The female head of the household will be followed because it is expected that she will be the household member that i. is mainly responsible for drinking water management, and ii. is at home most of the day and thus making it logistically feasible to obtain spot urine samples throughout the study.

At monthly intervals, participating households will be visited to assess filter use using self report as well as objective indicators. Additionally, in each round of follow-up, drinking water samples will be taken in all participating households for both microbiological and arsenic testing. Additionally, the female head of household will be invited to provide spot urine samples for total urinary arsenic at each round of follow up.

For arsenic testing samples of stored drinking water will be collected and analysed for total arsenic. Additionally, in intervention households, samples of source water will also be collected to assess the percentage removal of Arsenic by the Pureit AS+ filter. Water samples will be collected in polyethylene bottles pre-washed with nitric acid water and nitric acid (0.1% v/v) will be added after collection at the laboratory as a preservative (Roychowdhury, 2008). Samples will be stored in ice box until arrival to the lab and stored at 4°C until shipment to the laboratory for analysis. Total water arsenic will be measured by Flow Injection Hydride Generation Atomic Absorption Spectrometry (FI-HG-AAS) and or Inductively coupled plasma mass spectrometry (ICP-MS).

For microbiological testing, in each round of follow-up, in intervention households water samples will be collected of i. stored drinking water (whether this is from the intervention filter or another container), ii. in a 25% random sample, samples will also be taken of influent water (source water) and effluent water out of the filter (if they keep their drinking water elsewhere). For control households, water samples will be collected of i. stored drinking water and, ii. in a 25% random sample, from the water source. Untreated drinking water will be collected to determine technology performance by comparing effluent and influent water quality. For the stored drinking water, the householder will be asked if there is any drinking water in the house at that moment and a sample will be collected from the vessel that the householder identifies as being the main container used at that moment to fill a cup or glass for drinking. All samples for microbial analysis will be collected in sterile Whirl-Pak™ bags containing a tablet of sodium thiosulfate to neutralize any disinfectant. Samples will be placed on ice and processed within 4-6 hours of collection to assess TTC levels. Microbiological assessment will be performed using a DelAgua field incubator (University of Surrey) in accordance with Standard Methods (Eaton et al., 2005).

Acceptability and major limitations with the filtration technology will be assessed during the final follow-up visit. The acceptability of the technology will be evaluated by conducting household surveys, in-depth interviews (IDI) and focus group discussions (FGDs). A subsample of male and female heads of households will be asked to participate in FGDs at the end of the study to provide feedback on the technology including perceived benefits and limitations.

ELIGIBILITY:
Households will be eligible to participate in the study if (i) the water identified as drinking during the baseline survey has an arsenic concentration that exceeds 50 µg/L, when measured using a rapid portable field testing kit, (ii) an alternative arsenic mitigation project is not underway for the household at the time of enrolment, (iii) the household is within the designated geographical area of the study, (iv) the household lives permanently in the area and anticipates living in the area for the next 6 months, (v) the household is willing to participate and (vi) the female head of the household is at least 18 years, is able to provide consent (has no cognitive impairments) and accepts to provide urine samples.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total urinary arsenic | 4 months
  To assess the effectiveness of the Unilever Pureit As+ technology in decreasing the body burden of arsenic, measured in terms of total urinary arsenic

SECONDARY OUTCOMES:
Total arsenic removal in drinking water | 4 months
  Median and arithmetic mean of total arsenic concentration in intervention vs. control households stored drinking water
Total arsenic reduction in filtered water | 4 months
  To assess total arsenic removal performance in drinking water of the Unilever Pureit As+ technology in the field (Mean % removal).
Mean TTC reduction in drinking water | 4 months
  Williams mean of CFU/100 mL in intervention vs. control household stored drinking water
Self-reported use of the intervention | 4 months
  To examine consistent use of Unilever Pureit As+ technology, for children <5 years and all household members
Consistent use | 4 months
  To examine consistent use of Unilever Pureit As+ technology using objective indicators of use
Prevalence of diarrhoea among <5s | 4 months
  To examine the impact of the Unilever Pureit As+ technology on reported diarrhoea among children under 5 years
Prevalence of diarrhoea among all family members | 4 months
  5) To examine the impact of the Unilever Pureit As+ technology on reported diarrhoea among all family members.
Bacterial removal | 4 months
  Mean % removal (log reduction) of TTC for intervention households

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clasen, JD MSc PhD, Principal Investigator — LSHTM & Emory University
Locations (1):
- Gobardanga Seba Farmer's Samity (GSFS), Gobardanga, North 24 Parganas, West Bengal, India